CLINICAL TRIAL: NCT04920279
Title: Validity Of The Turkish Version Of Activities-Specific Balance Confidence Scale In Patients With Diabetes Mellitus
Brief Title: Validity Of Turkish Version Of ABC Scale In Diabetes Mellitus Patients
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Feride Sabırlı, Researcher, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Other Study IDs: IstPMRTRH-FS
Record Dates: First submitted 2021-06-03; First posted 2021-06-09 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus; Balance; Distorted; Evaluations, Diagnostic Self
Keywords: balance; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The patients with diabetes mellitus: When patients with diabetes mellitus admitted to our outpatient clinic if they have inclusion criteria, we have used the ABC questionnaire. And we have done perform Time Up And Go Test twice respectively.

SUMMARY:
Activities-specific Balance Confidence (ABC) scale is a well-known tool to evaluate functional balance. Diabetic patients suffer more often from balance disorders than the rest of the population. The aim is to investigate the validity of the Turkish version of ABC short form in patients with diabetes mellitus (DM).

DETAILED DESCRIPTION:
Thirty patients with DM will be included according to the inclusion and exclusion criteria. All the participants will be evaluated by ABC form and Timed Up and Go Test (TUG). The Cumulative Illness Rating Scale (CIRS ) will be used for all the patients.

ABC scale is a self-assessment test with 16 items that helps assess balance impairments and falling risk, and it also investigates how confident people are while they are in some specific activities both indoors, and outdoors. Total score changes between 0-100.

The HbA1c values of all patients will be noted if a blood test will be performed in the last three months.

ELIGIBILITY:
Inclusion Criteria:

* 45-75 years old
* Diabetes mellitus
* The complete existence of the data to be used in the study in the records of our hospital

Exclusion Criteria:

* Not having any other additional disease that will affect balance coordination
* No lower extremity joint replacement or lower extremity amputation at any level

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Validity of the Turkish Version of Activities-specific Balance Confidence Scale in Patients With Diagnosis of the Diabetes Mellitus Before. | A single point in time (1 day)
  The Activities-specific Balance Confidence Scale (ABC Scale) is a structured questionnaire that measures an individual's confidence in performing activities without losing balance. Total score ranges from 0% to 100%. Lower than 50 %: low level; 50-80 %: moderate level above 80 %: high level of physical functioning

CONTACTS AND LOCATIONS:
Overall Officials: Nurdan Paker, Prof, Principal Investigator — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Physical Medicine Rehabilitation Training & Research Hospital, Istanbul
  - IstanbulPMRTRH, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Powell LE, Myers AM. The Activities-specific Balance Confidence (ABC) Scale. J Gerontol A Biol Sci Med Sci. 1995 Jan;50A(1):M28-34. doi: 10.1093/gerona/50a.1.m28. PMID 7814786
- [Background] Sprint G, Cook DJ, Weeks DL. Toward Automating Clinical Assessments: A Survey of the Timed Up and Go. IEEE Rev Biomed Eng. 2015;8:64-77. doi: 10.1109/RBME.2015.2390646. Epub 2015 Jan 12. PMID 25594979
- [Background] Miller MD, Paradis CF, Houck PR, Mazumdar S, Stack JA, Rifai AH, Mulsant B, Reynolds CF 3rd. Rating chronic medical illness burden in geropsychiatric practice and research: application of the Cumulative Illness Rating Scale. Psychiatry Res. 1992 Mar;41(3):237-48. doi: 10.1016/0165-1781(92)90005-n. PMID 1594710
- [Background] Paker N, Bugdayci D, Demircioglu UB, Sabirli F, Ozel S. Reliability and validity of the Turkish version of Activities-specific Balance Confidence scale in symptomatic knee osteoarthritis. J Back Musculoskelet Rehabil. 2017;30(3):461-466. doi: 10.3233/BMR-150335. PMID 27858674